CLINICAL TRIAL: NCT00460460
Title: A Phase I, Open-label, Dose Escalation Study to Assess the Safety, Tolerability & Pharmacokinetics of AZD4877 Administered Once Weekly in Adult Patients With Recurrent or Refractory AML, PH Negative ALL, NHL or MN
Brief Title: Phase I, Open-label, Dose Escalation of AZD4877 in Hematologic Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated due to low enrollment
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D2782C00002
Record Dates: First submitted 2007-04-12; First posted 2007-04-16 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Lymphoma
Keywords: Phase I; cancer; lymphoma; leukemia; myeloma; AML; ALL; NHL; MM
MeSH Terms: conditions — Lymphoma; Neoplasms; Leukemia; Neoplasms, Plasma Cell | interventions — N-(3-aminopropyl)-N-(1-(5-benzyl-3-methyl-4-oxo-(1,2)thiazolo(5,4-d)pyrimidin-6-yl)-2-methylpropyl)-4-methylbenzamide

INTERVENTIONS:
Drug: AZD4877

SUMMARY:
The primary purpose of this study is to find out what the maximum tolerated dose is for an experimental drug called AZD4877 based on the side effects experienced by patients that receive AZD4877 on a weekly basis in these diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML, a certain type of ALL, NHL and MM
* certain types of cancer of the lymph nodes
* certain types of leukemias (blood cancers)
* disease has or will fail with other treatments
* relatively good overall health other than your cancer

Exclusion Criteria:

* poor bone marrow function (not producing enough blood cells)
* serious heart conditions
* poor liver or kidney function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2007-03; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Ochs, MD, Study Director — AstraZeneca
Locations (3):
- United States (2):
  - Research site, Buffalo, New York
  - Research Site, New York, New York
- Research Site, Toronto, Ontario, Canada